CLINICAL TRIAL: NCT04936997
Title: Immune Response to the COVID-19 Vaccine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012325795-B
Record Dates: First submitted 2021-06-18; First posted 2021-06-23 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Covid19; Cancer; Malignancy; Vaccine Response Impaired
Keywords: Covid-19 vaccine; Pfizer Covid-a9 vaccine; Covid vaccine study
MeSH Terms: conditions — COVID-19; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 3rd COVID-19 vaccine (2nd booster) (Experimental): Patients who were a part of the non-interventional portion of the study are eligible to receive a third COVID-19 Pfizer vaccine.
  Interventions: Biological: SARS-COV2 Pfizer Vaccine

INTERVENTIONS:
Biological: SARS-COV2 Pfizer Vaccine — Vaccine for the prevention of coronavirus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).

SUMMARY:
Explore the effects on immune response to include a potential third vaccine for the cancer cohort.

DETAILED DESCRIPTION:
In recent work performed by the University of Arizona Cancer Center team, 59 patients with a known diagnosis of a solid tumor malignancy on active immunosuppressive cancer therapy were enrolled through the University of Arizona Cancer Center during their routine care. These subjects had a decreased response with the vaccine when compared to the health cohort. The investigators are amending this study to explore the effects on immune response to include a potential third vaccine for the cancer cohort. This will increase the visits required to approximately two more visits. It will require two additional blood samples, one 48 hours prior to third vaccine and the second, 5-11 days after the third vaccine. The following protocol will be for the subjects that decide to continue onto a third vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have active solid tumor malignancy diagnosis
2. On active chemotherapy
3. Received two prior SARS-COV2 Pfizer vaccines
4. Age ≥ 18 years
5. Ability to understand and the willingness to sign a written informed consent
6. Agree to comply with study procedures
7. Subjects previously enrolled under the main study

Exclusion Criteria:

1. History of HIV or organ/bone marrow transplant
2. Actively receiving immunotherapy
3. On active, chronic immunosuppression (>10 mg daily dose of prednisone equivalent)
4. Currently incarcerated or residence of another state
5. Speaks a language other than English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2022-05-08 (Actual)

PRIMARY OUTCOMES:
Immune response | 3 months
  Evaluating immune response to a second COVID-19 vaccination booster (3rd vaccine) in patients with solid tumor malignancies on immunosuppressive cancer therapies by antibody quantification in blood samples.

SECONDARY OUTCOMES:
Adverse events | 3 months
  Evaluating immune response to a second COVID-19 vaccination booster (3rd vaccine) in patients with solid tumor malignancies on immunosuppressive cancer therapies by T-cell quantification in blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Rachna Shroff, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Derived] Shroff RT, Chalasani P, Wei R, Pennington D, Quirk G, Schoenle MV, Peyton KL, Uhrlaub JL, Ripperger TJ, Jergovic M, Dalgai S, Wolf A, Whitmer R, Hammad H, Carrier A, Scott AJ, Nikolich-Zugich J, Worobey M, Sprissler R, Dake M, LaFleur BJ, Bhattacharya D. Immune responses to two and three doses of the BNT162b2 mRNA vaccine in adults with solid tumors. Nat Med. 2021 Nov;27(11):2002-2011. doi: 10.1038/s41591-021-01542-z. Epub 2021 Sep 30. PMID 34594036